CLINICAL TRIAL: NCT05297539
Title: Optimization of the Role of Action Observation in the Post-operative Rehabilitation of the Total Knee Prosthesis
Brief Title: Optimization of the Role of Action Observation in the Post-operative Rehabilitation of the Total Knee Prosthesis: (LOARAL 2)
Acronym: LOARAL 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-A03000-41
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Knee Surgery; Rehabilitation; Point Light Display

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): Control group who will do usual rehabilitation + visualization of videos representing monuments + a 3-meter round-trip walk
- Experimental group 1 (Experimental): Experimental group 1 who will do usual rehabilitation + visualization of non focused point-light human actions + a 3-meter round-trip walk
  Interventions: Other: Point light display
- Experimental group 2 (Experimental): Experimental group 2 who will do usual rehabilitation + visualization of focused point-light human actions + a 3-meter round-trip walk
  Interventions: Other: Point light display

INTERVENTIONS:
Other: Point light display — Visualization of point-light human actions
  Arms: Experimental group 1; Experimental group 2

SUMMARY:
The LOARAL 2 project concerns patients who have undergone total knee arthroplasty to treat symptomatic osteoarthritis. Patient will be divided into three groups: a control group where patients will do standard rehabilitation associated with the judgments of videos represented non-human action and two experimental groups where patients will do standard rehabilitation associated with the judgement of human point-light display. The aim of this study is to measure the benefits of attentional focus and sex correspondence in the use of point-light display for the rehabilitation of patients with a total arthroplasty of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers over 18 years of age who have undergone knee surgery

Exclusion Criteria:

* Any locomotor condition not due to knee surgery
* Uncorrected visual disturbances
* Comorbidity altering locomotion (history of stroke, neurological condition, inflammatory rheumatism)

Non randomization criteria:

* Cognitive disorders (Mini Mental State Examination <21)
* Depressive disorders (Beck Inventory index> 9)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
The score obtained on the Western Ontario and McMaster (WOMAC) test at inclusion and at the end of the program. | Rehabilitation during 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No